CLINICAL TRIAL: NCT02362659
Title: Antithrombotic Strategy Variability In ATrial Fibrillation and Obstructive Coronary Disease Revascularized With PCI
Brief Title: Antithrombotic Strategy Variability In ATrial Fibrillation and Obstructive Coronary Disease Revascularized With PCI - The AVIATOR 2 Registry
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: GCO 14-1543-00002; CV185-376 (Other: BMS); PD14-03987 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: non-valvular; atrial fibrillation; percutaneous coronary intervention
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Antiplatelet agent plus anticoagulant: an antithrombotic regimen comprising one single antiplatelet agent plus an anticoagulant
- DAPT alone: an antithrombotic regimen consisting of dual antiplatelet therapy (DAPT) alone
- DAPT plus anticoagulant: an antithrombotic regimen consisting of DAPT plus anticoagulant therapy

SUMMARY:
The purpose of this observational registry was to compare the safety and efficacy of an antithrombotic regimen comprising one single antiplatelet agent plus an oral anti-thrombotic versus those consisting of DAPT alone or DAPT plus oral antithrombotic therapy. This registry assessed whether the antithrombotic therapy intensity would vary positively with physician perceived ischemic risk at the time of percutaneous coronary intervention (PCI), and whether an inverse association would be observed with perceived bleeding risk.

This study also evaluated the physician use of objective benefit-risk assessment scores and their influence on prescription of antithrombotic therapy in atrial fibrillation (AF) patients undergoing PCI. Additionally the study investigated whether patient perceived relevance and accessibility of anti-platelet and anticoagulant treatment regiments would predict treatment adherence and whether non-adherence would independently influence outcome.

Approximately 514 subjects with non-valvular AF undergoing all-comer PCI were enrolled at 11 sites in North America and Europe. Follow-up was done via telephone by trained research coordinators at each participating site at 30 days, 6 months and 12 months.

DETAILED DESCRIPTION:
The current AHA guidelines on AF for patients undergoing PCI are non-specific as they recommend "low-dose aspirin (less than 100 mg per d) and/or clopidogrel (75 mg per d), which may be given concurrently with anticoagulation to prevent myocardial ischemic events, but these strategies have not been thoroughly evaluated and are associated with an increased risk of bleeding.

Finding the right balance that minimizes bleeding risk and maintains anti-ischemic efficacy remains a complex and controversial clinical dilemma in these unique patients. The arrival of novel antiplatelet agents and antithrombotics on the scene has led to an exponential increase in the combinations that may be employed by clinicians in real-life situations. The sheer number of combinations means that the best APT and OAC combination based on RCT data will not be known for many years. It has therefore become imperative that the investigators strive to create better methods to gauge the comparative safety and efficacy for various antiplatelet and antithrombotic combination strategies in AF patients undergoing PCI. To the best of the investigators knowledge, no contemporary prospective registry of real-life patients with AF undergoing PCI exists or has been initiated to date. Additionally, the factors influencing physician choice of treatment strategy as well as factors predicting patient adherence in this population is largely unknown.

This is a multi-center, multinational, observational prospective registry prospective analysis of 514 patients with non-valvular AF undergoing all-comer PCI at 11 Northern American and European centers. Patients were followed for 12 months. Data was collected prospectively. All-antiplatelet and anti-thrombotic treatment regimen were at the physicians' discretion. The investigators studied various combinations of antiplatelet and antithrombotic therapies, characterized the bleeding and ischemic risk in patients with atrial fibrillation undergoing PCI and determined physician and patient centered factors influencing prescription patterns and patient adherence.

Patients with non-valvular atrial fibrillation who have undergone successful PCI were enrolled as soon as possible post procedure and no later than before discharge of the index admission. The treating physician (interventional or non-interventional cardiologist) that prescribed the anti-platelet or/and anticoagulant therapy also completed the physician questionnaire. A different, patient centered questionnaire was completed by the patient. The Principal Investigator or designee provided instructions to enrolled subjects and physicians on how to use the hand held electronic device or how to complete the paper questionnaire and clarify any questions about the questionnaires. The enrolled subjects and physicians themselves entered the responses to the questionnaire on the electronic hand held device or the paper questionnaire. Only patients with completed questionnaires were considered enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-valvular atrial fibrillation during hospitalization.
* Preexisting atrial fibrillation.
* Successful all-comer percutaneous coronary intervention:

Procedural success is defined as a reduction of residual luminal diameter stenosis to <50% without in-hospital death, AMI or the need for emergency CABG.

* Over 18 years of age
* Able to provide written informed consent

Exclusion Criteria:

* Atrial fibrillation due to reversible causes (e.g., thyrotoxicosis, pericarditis)
* Valvular atrial fibrillation secondary to severe mitral stenosis or prosthetic heart valve
* Women who are of childbearing potential Treatment with other investigational drugs or devices within 30 days before enrolment or planned use of investigational drugs or devices during the study
* Life expectancy <12 months due to non-cardiac comorbidities
* Active alcohol, drug abuse, psychosocial reasons making study participation impractical
* Severe renal insufficiency (calculated creatinine clearance < 30 mL/min) or dialysis
* Clinically overt stroke within the last 3 months
* Known hypersensitivity or contraindication to aspirin, clopidogrel, prasugrel, ticagrelor, dabigatran, rivaroxaban, apixaban, edoxaban or warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 514 patients with non-valvular AF undergoing all-comer PCI at 11 Northern American and European hospital centers.
Sampling Method: Non-Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 months
  Efficacy as measured by composite of All-cause death, non-fatal MI, stroke, stent thrombosis, clinically driven target lesion revascularization at 1 year - MACCE (major adverse cardiovascular and cerebrovascular events)
bleeding risk | 12 months
  Safety as measured by bleeding according to the Bleeding Academic Research Consortium (BARC) bleeding definitions (BARC 2,3 or 5)

SECONDARY OUTCOMES:
Net adverse clinical events | 12 months
  Net adverse clinical events (NACE) - composite occurrence of all MACCE and major bleeding.
Association between subjective and objective measures of ischemic and bleeding risk | 12 months
  Ischemic events assessed by CHADS, CHA2DS2-VASc is a non-valvular AF thromboembolism risk score.
Modes of antithrombotic therapy cessation | 12 months
  Modes of antiplatelet and antithrombotic therapy cessation: discontinuation (physician recommended), interruption (e.g. for surgery/procedures), disruption (non-recommended)

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Usman Baber, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Chandrasekhar J, Mastoris I, Baber U, Sartori S, Schoos M, Bansilal S, Dangas G, Mehran R. Antithrombotic strategy variability in ATrial fibrillation and obstructive coronary disease revascularized with PCI-rationale and study design of the prospective observational multicenter AVIATOR 2 registry. Am Heart J. 2015 Dec;170(6):1234-42. doi: 10.1016/j.ahj.2015.08.023. Epub 2015 Sep 21. PMID 26678646
- [Derived] Chandrasekhar J, Baber U, Sartori S, Goel R, Nicolas J, Vogel B, Snyder C, Kini A, Briguori C, Witzenbichler B, Iakovou I, Sardella G, Marzo K, DeFranco A, Stuckey T, Chieffo A, Colombo A, Shlofmitz R, Capodanno D, Dangas G, Pocock S, Mehran R. Antithrombotic strategy variability in atrial fibrillation and obstructive coronary disease revascularised with percutaneous coronary intervention: primary results from the AVIATOR 2 international registry. EuroIntervention. 2022 Oct 7;18(8):e656-e665. doi: 10.4244/EIJ-D-21-01044. PMID 35656720